CLINICAL TRIAL: NCT01026298
Title: The Relationship Between Asthma and Obstructive Sleep Apnea (OSA) - A Pilot Study of the Effects of OSA and Its Treatment on Asthma
Brief Title: Asthma and Obstructive Sleep Apnea (OSA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2012-1038; H-2007-0034 (Other: HS IRB); A534285 (Other: UW, Madison); SMPH/MEDICINE/PULMON MED (Other: UW, Madison)
Record Dates: First submitted 2009-12-02; First posted 2009-12-04 (Estimated); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: Asthma; Obstructive Sleep Apnea
Keywords: asthma; obstructive sleep apnea; severe asthma; OSA
MeSH Terms: conditions — Asthma; Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (No Intervention): 8 weeks, no intervention for OSA
- CPAP group (Active Comparator): 8-week randomized-controlled period of CPAP treatment
  Interventions: Other: FDA-Approved Treatment

INTERVENTIONS:
Other: FDA-Approved Treatment — 8 weeks of treatment with Continuous Positive Airway Pressure (CPAP)
  Arms: CPAP group

SUMMARY:
Obstructive sleep apnea (OSA) is a common but under-diagnosed form of sleep disordered breathing (SDB). Asthma is a common disease with rising prevalence, which continues to pose significant morbidity and costs. In spite of considerable progress in our understanding of asthma, a large number of individuals with asthma continue to have symptoms and subsequently, have a poor functional status, poor quality of life and increased health care costs. In many cases no apparent cause is found and optimal therapy does not achieve its goal. While recent data suggests that OSA is common in severe asthma, the prevalence of OSA and its predisposing factors have not been studied.

ELIGIBILITY:
Inclusion Criteria:

* presence of not well-controlled (NWC) asthma (National Asthma Education and Prevention Program Guidelines step 2, 3, 4), as diagnosed by an asthma physician
* stable doses of standard therapy for 2 months prior to enrollment. These regimens will include: inhaled corticosteroids (ICS) for mild-persistent step; ICS and inhaled long-acting β-adrenergics (LABA) or ICS and leukotriene modifier (LTMs) agents for moderate-persistent step; high doses of ICS, LABA or LTMs, with or without oral steroids at stable doses, for patients in severe step
* adherence to the current asthma medications regimen, demonstration of a proper inhaler technique; agreement for maintaining the same asthma regimen (except rescue bronchodilators) as clinical condition permits (if an exacerbation occurs during the first 4-week period, the subject will be excluded as discussed below), and willingness to complete diaries of asthma symptoms, rescue bronchodilator use, peak flow meter (PEF) recordings as well as asthma-related urgent doctor's and emergency room visits and hospitalizations for the 3 months duration of the study
* moderate to high probability for OSA (SA-SDQ scores ≥31 for males and ≥28 for females) or high clinical suspicion for OSA
* preliminary agreement to treatment with continuous positive airway pressure (CPAP) if OSA is identified and current CPAP treatment criteria are met [patients with moderate to severe OSA (AHI>15 events/hour), patients with mild OSA (AHI 5-15 events/hour) in association with EDS or co-morbid conditions (HTN, stable ischemic heart disease, prior stroke, impaired cognition, mood disorders, insomnia
* ability to read and write
* ability and willingness to return to the Medical Center as required by the study protocol.

Exclusion Criteria:

* asthma exacerbation in the prior 2 months
* acute sinusitis
* poorly controlled rhinitis or gastroesophageal reflux disease (GERD)
* any unstable medical or psychiatric illness likely to impede participation in the protocol during the next year
* evidence of co-existent lung disease, in particular allergic broncho-pulmonary aspergillosis or chronic obstructive pulmonary disease (COPD)
* treated OSA or another primary sleep disorder
* evidence of medical instability due to OSA at first sleep study visit
* subjects with excessive daytime sleepiness to a degree that puts the subject or people around at risk of accidents (motor vehicle or work-related). In these cases we will facilitate expedited sleep evaluations through primary providers
* historical evidence of collagen vascular disease
* craniofacial abnormalities precluding the use of CPAP; 11) current cigarette smoking or within the prior 6 months (self-report and medical records
* pregnancy (documented via urine-human chorionic gonadotropin detection test) or desire to become pregnant during the following 3 months
* mental impairment limiting the ability to provide informed consent
* current alcohol (as per the NIH cutoffs56 presented below) or recreational drug use (for both, based on medical records review and self-report without any prospective recording); women drinking more than 3 drinks at one time or more than 7 standard drinks a week or men drinking more than 4 drinks at one time or more than 14 standard drinks a week will be excluded. A standard drink is defined as one can or bottle of beer (12 fl oz), one glass of wine (5 fl oz), or one mixed drink containing 1.5 fl oz of hard liquor.

Ages: 18 Years to 73 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 744 (Actual)
Dates: Start 2007-03 (Actual); Primary Completion 2012-05-07 (Actual); Study Completion 2012-06-25 (Actual)

PRIMARY OUTCOMES:
To determine the prevalence and risk factors for OSA symptoms in a specialty clinic-based sample of individuals with asthma. | 7 days

SECONDARY OUTCOMES:
To assess changes in subjective and objective asthma measures in subjects with asthma and co-morbid OSA, after 8 weeks of treatment with continuous positive airway pressure (CPAP) versus no intervention (control). | 56 days
To examine whether 8 weeks of CPAP for OSA improves quality of life, insomnia, daytime sleepiness and fatigue, and health resource utilization in individuals with asthma. | 56 days

CONTACTS AND LOCATIONS:
Overall Officials: Mihaela Teodorescu, MD, Principal Investigator — UW Madison
Locations (1):
- Univeristy of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No